CLINICAL TRIAL: NCT03223337
Title: A Phase 1, Open-label, Non-randomized, Parallel Group, Single-dose Adaptive Study in Adults With Hepatic Impairment and Matched, Healthy Control Participants With Normal Hepatic Function
Brief Title: Daprodustat Hepatic Impairment Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 200231
Record Dates: First submitted 2017-07-18; First posted 2017-07-21 (Actual); Results first posted 2019-09-04 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-08

CONDITIONS: Anaemia
Keywords: GSK1278863; Daprodustat; Healthy control; Single dose; Hepatic Impairment
MeSH Terms: conditions — Anemia | interventions — GSK1278863

STUDY DESIGN:
Intervention Model Description: All subjects will receive 6 mg of daprodustat as a single oral dose in parallel way throughout the study period.
Masking Description: This will be an open-label study and no blinding will be performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Subjects with moderate hepatic impairment: Part 1 (Experimental): Approximately 8 subjects with moderate hepatic impairment will receive 6 mg of daprodustat as a single oral dose in the fasted state. This group will include at least one subject with a Child-Pugh score of 7, one with a score of 8 and one with a score of 9. The group will also include at least one female and at least one male subject.
  Interventions: Drug: Daprodustat (GSK1278863)
- Matched Healthy controls: Part 1 (Active Comparator): Approximately 8 healthy controls, matched in gender, age and BMI to subjects with moderate hepatic impairment, will receive 6 mg of daprodustat as a single oral dose in the fasted state. The group will include at least one female and at least one male subject.
  Interventions: Drug: Daprodustat (GSK1278863)
- Subjects with either mild or severe hepatic impairment: Part 2 (Experimental): Approximately 8 subjects with mild or severe hepatic impairment will receive 6 mg of daprodustat as a single oral dose in the fasted state. This group will include at least one subject with a Child-Pugh score of 5 and one with a score of 6 for mild hepatic impairment and at least one subject with a Child-Pugh score of 10 or 11 and one with a score of 12 or 13 for severe hepatic impairment. The group will also include at least one female and at least one male subject.
  Interventions: Drug: Daprodustat (GSK1278863)
- Matched healthy controls: Part 2 (Active Comparator): Approximately 8 healthy controls, matched in gender, age and BMI to subjects with mild or severe hepatic impairment, will receive 6 mg of daprodustat as a single oral dose in the fasted state. The group will include at least one female and at least one male subject.
  Interventions: Drug: Daprodustat (GSK1278863)

INTERVENTIONS:
Drug: Daprodustat (GSK1278863) — Daprodustat (GSK1278863) 6 mg tablet will be given to all subjects as a single dose via oral route. Daprodustat (GSK1278863) is a 9.0 millimeter (mm) round, compound radius, white film coated tablet.

SUMMARY:
Daprodustat (GSK1278863), is a small molecule currently in development for the treatment of anemia of chronic kidney disease (CKD). Results of the earlier studies shows that liver is involved in the clearance of Daprodustat and hence, hepatic impairment can affect Daprodustat levels in the body. This single dose study will assess the effect of liver impairment on the pharmacokinetics (PK) and pharmacodynamics (PD) of daprodustat. The study will be conducted in two parts, Part 1 will include subjects with moderate hepatic impairment and matched healthy control subjects whereas Part 2 will include subjects will either mild or severe hepatic impairment and matched healthy control subjects. Approximately 8 subjects will be included in each of the group and all subjects will receive 6 milligram (mg) of daprodustat as a single oral dose in the fasted state. Total duration of participation in the study for a subject will be up to 7 weeks.

ELIGIBILITY:
Inclusion Criteria:

For all subjects:

* Subject must be at least 18 years of age inclusive, at the time of signing the informed consent.
* Hemoglobin values at screening <=16.0 gram per deciliter (g/dL) for males and <=14.0 g/dL for females.
* Body weight >=45 kilograms (kg) and body mass index (BMI) within the range 18-40 kg per meter square (kg/m^2) (inclusive).
* Male or female subjects will be included. A female subject is eligible to participate if she is not breastfeeding, and at least one of the following applies: Not pregnant as confirmed by two pregnancy tests; Not a woman of childbearing potential (WOCBP); For WOCBP that are currently utilizing a highly-effective contraceptive method prior to enrolment, agrees to follow the contraceptive guidance during the treatment period to the follow-up visit.
* Capable of giving signed informed consent form.

Additional inclusion criteria for Hepatically-Impaired subjects:

* Subjects in Part 1 with Moderate Hepatic Impairment Only (Cohort 1): Is considered to have moderate hepatic impairment (of any etiology) and has been clinically stable for at least 1 month prior to screening. To be classified as having moderate hepatic impairment, subjects must have a Child-Pugh (Class B) score of 7-9 AND previous confirmation of liver cirrhosis by liver biopsy or other medical imaging technique (including laparoscopy, computerized tomography (CT) scan, magnetic resonance imaging (MRI) or ultrasonography) associated with an unambiguous medical history (such as evidence of portal hypertension).
* Subjects in Part 2 with Mild OR Severe Hepatic Impairment Only (Cohort 3; if conducted): Is considered to have mild or severe hepatic impairment (of any etiology) and has been clinically stable for at least 1 month prior to screening. To be classified as having mild OR severe hepatic impairment, subjects must have: classified as having mild hepatic impairment, subjects must have a Child- Pugh (Class A) score of 5-6 AND previous confirmation of chronic liver disease by liver biopsy or other medical imaging technique (including laparoscopy, CT scan, MRI or ultrasonography) associated with an unambiguous medical history (such as evidence of portal hypertension); classified as having severe hepatic impairment, subjects must have Child- Pugh (Class C) score of 10-13 AND previous confirmation of chronic liver disease by liver biopsy or other medical imaging technique (including laparoscopy, CT scan, MRI or ultrasonography) associated with an unambiguous medical history (such as evidence of portal hypertension).
* Supplemental inclusion criteria for ALL hepatically-impaired subjects: Chronic (>6 months), stable (no acute episodes of illness due to deterioration in hepatic function within the previous 1 month prior to screening) hepatic impairment due to any etiology. Subjects must also remain stable throughout the Screening period. Assessment of the stability of the subjects hepatic function will be determined by the investigator.

Additional inclusion criteria for healthy control subjects:

* Healthy control subjects will be matched for age +/-10 years to subjects in the respective hepatic impairment cohort but must also be at least 18 years of age inclusive, at the time of signing the informed consent.
* Healthy as determined by the investigator or medically qualified designee based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring.
* A subject with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied may be included only if the investigator and/or the Medical Monitor agree and document that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Healthy control subjects will be matched for BMI +/-15% to subjects in the respective hepatic impairment cohort but must also remain in the range of body weight >=45 kg and BMI within the range 18-38 kg/m^2 (inclusive).

Exclusion Criteria:

For all subjects:

* QT interval corrected for heart rate according to Fridericia's formula (QTcF) >500 milliseconds (msec).
* Recent history of deep vein thrombosis, pulmonary embolism or other thrombosis related condition. Any prior medical history in these areas will be reviewed and approved by the PI and the sponsor's Medical Monitor on a case by case basis as needed.
* Myocardial infarction or acute coronary syndrome, stroke or transient ischemic attack within the 12 weeks prior to enrollment.
* Subjects with a pre-existing condition (other than liver disease) interfering with normal gastrointestinal anatomy or motility that could interfere with the absorption, metabolism, and/or excretion of daprodustat.
* Subjects that have undergone cholecystectomy within the past 3 months.
* Subjects with chronic inflammatory joint disease (example, scleroderma, systemic lupus erythematosis, rheumatoid arthritis).
* History of malignancy within the prior 2 years or known kidney mass >3 centimeter (cm) (end stage renal disease subjects with impairment only) OR currently receiving treatment for cancer. ONLY exception is localized squamous cell or basal cell carcinoma of the skin definitively treated 12 weeks prior to enrollment.
* Class IV heart failure, as defined by the New York Heart Association (NYHA) functional classification system.
* Current enrolment or past participation (i.e., administration of last dose of investigational study treatment) within the last 30 days (or 5 half-lives, whichever is longer) before Day 1 in this or any other clinical study involving an investigational study treatment or any other type of medical research.

Exclusion criteria for Hepatically-Impaired subjects:

* Present of 8 times Upper limit of normal (ULN) elevations in Aspartate aminotransferase (AST), Alanine aminotransferase (ALT), or bilirubin.
* Subjects with any other medical condition which, in the judgment of the investigator and Medical Monitor, could jeopardize the integrity of the data derived from that subject or the safety of the subject.
* Subjects with advanced ascites (Grade 3).
* Subjects with refractory encephalopathy as judged by the investigator or significant Central Nervous System (CNS) disease (example dementia, or seizures) which the investigator considers will interfere with the informed consent, conduct, completion, or results of this trial or constitutes an unacceptable risk to the subject.
* Subjects with functional Transjugular Intrahepatic Portosystemic Shunt (TIPS) placement.
* Presence of hepatopulmonary or hepatorenal syndrome.
* Presence of primarily cholestatic liver diseases.
* History of liver transplantation.
* Subjects with signs of active infection, including active spontaneous bacterial peritonitis.
* Subjects with unstable cardiac function or subjects with hypertension whose blood pressure is not controlled (based on the investigator's discretion).
* Diabetic subjects whose diabetes is not controlled (based on the investigator's discretion).

Exclusion criteria for healthy control subjects:

* Exposure to more than 4 new chemical entities within 12 months prior to the first dosing day.
* Presence of Hepatitis B surface antigen (HBsAg) at screening or Positive Hepatitis C antibody test result at screening or within 3 months before the first dose of study treatment.
* Positive pre-study drug/alcohol screen.
* Positive human immunodeficiency virus (HIV) antibody test.
* Regular use of known drugs of abuse.
* Regular alcohol consumption within 6 months prior to the study defined as an average weekly intake of >14 drinks. One drink is equivalent to 12 g of alcohol: 12 ounces (360 mL) of beer, 5 ounces (150 mL) of wine or 1.5 ounces (45 mL) of 80 proof distilled spirits. One unit is equivalent to 8 g of alcohol: a half-pint (approximately 240 mL) of beer, 1 glass (125 mL) of wine or 1 (25 mL) measure of spirits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2017-07-24 (Actual); Primary Completion 2018-08-20 (Actual); Study Completion 2018-08-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- United States (2):
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Orlando, Florida

REFERENCES:
- [Derived] Mahar KM, Shaddinger BC, Ramanjineyulu B, Andrews S, Caltabiano S, Lindsay AC, Cobitz AR. Pharmacokinetics of Daprodustat and Metabolites in Individuals with Normal and Impaired Hepatic Function. Clin Pharmacol Drug Dev. 2022 May;11(5):562-575. doi: 10.1002/cpdd.1090. Epub 2022 Mar 30. PMID 35355447

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a two part study in adults with moderate (Part 1) and potentially mild (Part 2) hepatic impairment and matched, healthy control participants with normal hepatic function. This study was conducted at two centers in the United States of America (USA).
Pre-assignment Details: All participants received 6 milligrams (mg) of daprodustat (GSK1278863) as a single oral dose in the fasted state. A total number of 16 participants were enrolled in Part 1 and 21 participants were enrolled in Part 2 of the study. In total 37 participants were enrolled in the study.
Groups:
- Part 1: Moderate Hepatic Impairment Participants: Participants with moderate hepatic impairment received 6 mg of GSK1278863 as a single oral dose tablet in the fasted state during Part 1 of the study. This group included at least one participant with a Child-Pugh score of 7, 8 and 9 for moderate hepatic impairment.
- Part 1: Healthy Participants: Healthy control participants, matched to moderate hepatic impairment participants in gender, age and Body mass index (BMI) received 6 mg of GSK1278863 as a single oral dose tablet in the fasted state.
- Part 2: Mild Hepatic Impairment Participants: Participants with mild hepatic impairment received 6 mg of GSK1278863 as a single oral dose tablet in the fasted state during part 2 of the study. This group included at least one participant with a Child-Pugh score of 5 and 6 for mild hepatic impairment.
- Part 2: Healthy Participants: Healthy control participants, matched to mild hepatic impairment participants in gender, age and BMI received 6 mg of GSK1278863 as a single oral dose tablet in the fasted state in part 2 of the study.
Period: Part 1 (Up to 16 Days)
Arm/Group | Part 1: Moderate Hepatic Impairment Participants | Part 1: Healthy Participants | Part 2: Mild Hepatic Impairment Participants | Part 2: Healthy Participants
Started | 8 | 8 | 0 | 0
Completed | 8 | 8 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Part 2 (Up to 16 Days)
Arm/Group | Part 1: Moderate Hepatic Impairment Participants | Part 1: Healthy Participants | Part 2: Mild Hepatic Impairment Participants | Part 2: Healthy Participants
Started | 0 | 0 | 12 | 9
Completed | 0 | 0 | 12 | 9
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: Moderate Hepatic Impairment Participants | Part 1: Healthy Participants | Part 2: Mild Hepatic Impairment Participants | Part 2: Healthy Participants | Total
Number analyzed (Participants) | 8 | 8 | 12 | 9 | 37
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.5 (6.00) | 57.6 (7.15) | 61.9 (7.55) | 58.7 (8.03) | 59.7 (7.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2 | 2 | 6
  Male | 7 | 7 | 10 | 7 | 31
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  BLACK OR AFRICAN AMERICAN | 0 | 2 | 1 | 2 | 5
  WHITE - WHITE/CAUCASIAN/EUROPEAN HERITAGE | 8 | 6 | 6 | 6 | 26
  ASIAN - EAST ASIAN HERITAGE | 0 | 0 | 1 | 0 | 1
  WHITE - ARABIC/NORTH AFRICAN HERITAGE | 0 | 0 | 4 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Area Under the Concentration-time Curve From Time Zero (Pre-dose) Extrapolated to Infinite Time (AUC [0-infinity]) of GSK1278863 and Its Metabolites
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK1278863 and its metabolites; GSK2391220 (M2), GSK2506104 (M3), GSK2487818 (M4), GSK2506102 (M5), GSK2531398 (M6), and GSK2531401 (M13). Pharmacokinetic parameters were determined using standard non-compartmental methods. Pharmacokinetic Population comprised of all participants in the Safety Population for whom a pharmacokinetic sample was obtained and analyzed.
Time Frame: Pre-dose, 30 minutes, 1 hour, 1 hour 30 minutes, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 10 hours, 12 hours, 24 hours, 36 hours, 48 hours post-dose
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*nanogram per milliliter
Arm/Group | Part 1: Moderate Hepatic Impairment Participants | Part 1: Healthy Participants
Number analyzed (Participants) | 8 | 8
Hour*nanogram per milliliter
  GSK1278863 | 296.2407 (111.1) | 148.3225 (31.7)
  GSK2391220 (M2) | 77.6352 (56.9) | 47.1340 (30.9)
  GSK2487818 (M4) | 47.5557 (67.4) | 28.9896 (30.3)
  GSK2506102 (M5) | 16.8212 (43.9) | 11.2658 (29.4)
  GSK2506104 (M3) | NA (NA) — Data was not calculable for the metabolite GSK2506104 (M3) due to matrix-related suppression during the bio-analysis of the Part 1 pharmacokinetic plasma samples. | NA (NA) — Data was not calculable for the metabolite GSK2506104 (M3) due to matrix-related suppression during the bio-analysis of the Part 1 pharmacokinetic plasma samples.
  GSK2531398 (M6) | 33.9398 (49.2) | 20.9224 (27.7)
  GSK2531401 (M13) | 52.0606 (34.0) | 39.6044 (32.1)
Statistical Analysis 1: Comparison: Part 1: Moderate Hepatic Impairment Participants vs Part 1: Healthy Participants; Test type: Other; Ratio of Geometric Least Square(LS) Mean = 1.9973, 90% CI 2-sided [1.1063 to 3.6057] — Ratio of Geometric LS Mean for GSK1278863 (Moderate hepatic impairment participants versus Healthy participants) has been presented
Statistical Analysis 2: Comparison: Part 1: Moderate Hepatic Impairment Participants vs Part 1: Healthy Participants; Test type: Other; Ratio of Geometric LS Mean = 1.6471, 90% CI 2-sided [1.1267 to 2.4079] — Ratio of Geometric LS Mean for GSK2391220 (M2) (Moderate hepatic impairment participants versus Healthy participants) has been presented
Statistical Analysis 3: Comparison: Part 1: Moderate Hepatic Impairment Participants vs Part 1: Healthy Participants; Test type: Other; Ratio of Geometric LS Mean = 1.6404, 90% CI 2-sided [1.0744 to 2.5048] — Ratio of Geometric LS Mean for GSK2487818 (M4) (Moderate hepatic impairment participants versus Healthy participants) has been presented
Statistical Analysis 4: Comparison: Part 1: Moderate Hepatic Impairment Participants vs Part 1: Healthy Participants; Test type: Other; Ratio of Geometric LS Mean = 1.4931, 90% CI 2-sided [1.0876 to 2.0498] — Ratio of Geometric LS Mean for GSK2506102 (M5) (Moderate hepatic impairment participants versus Healthy participants) has been presented
Statistical Analysis 5: Comparison: Part 1: Moderate Hepatic Impairment Participants vs Part 1: Healthy Participants; Test type: Other; Ratio of Geometric LS Mean = 1.6222, 90% CI 2-sided [1.1594 to 2.2696] — Ratio of Geometric LS Mean for GSK2531398 (M6) (Moderate hepatic impairment participants versus Healthy participants) has been presented
Statistical Analysis 6: Comparison: Part 1: Moderate Hepatic Impairment Participants vs Part 1: Healthy Participants; Test type: Other; Ratio of Geometric LS Mean = 1.3145, 90% CI 2-sided [0.9896 to 1.7462] — Ratio of Geometric LS Mean for GSK2531401 (M13) (Moderate hepatic impairment participants versus Healthy participants) has been presented

2. Primary Outcome: Part 2: AUC (0-infinity) of GSK1278863 and Its Metabolites
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK1278863 and its metabolites; GSK2391220 (M2) , GSK2506104 (M3), GSK2487818 (M4), GSK2506102 (M5), GSK2531398 (M6), and GSK2531401 (M13). Pharmacokinetic parameters were determined using standard non-compartmental methods.
Time Frame: as for outcome 1
Population: Pharmacokinetic Population. Only those participants with data available at specified time point were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*nanogram per milliliter
Arm/Group | Part 2: Mild Hepatic Impairment Participants | Part 2: Healthy Participants
Number analyzed (Participants) | 8 | 7
Hour*nanogram per milliliter
  GSK1278863 | 299.8773 (39.9) | 205.7559 (37.2)
  GSK2391220 (M2) | 91.3799 (44.7) | 47.1647 (26.9)
  GSK2487818 (M4) | 63.6211 (40.1) | 31.7637 (28.4)
  GSK2506102 (M5) | 19.4020 (36.6) | 11.3374 (26.7)
  GSK2506104 (M3) | 91.7692 (41.0) | 50.1154 (28.3)
  GSK2531398 (M6) | 41.4666 (31.2) | 21.0066 (23.5)
  GSK2531401 (M13) | 46.7001 (66.5) | 31.9797 (40.9)
Statistical Analysis 1: Comparison: Part 2: Mild Hepatic Impairment Participants vs Part 2: Healthy Participants; Test type: Other; Ratio of Geometric LS Mean = 1.4574, 90% CI 2-sided [1.0350 to 2.0523] — Ratio of Geometric LS Mean for GSK1278863 (Mild hepatic impairment participants versus Healthy participants) has been presented
Statistical Analysis 2: Comparison: Part 2: Mild Hepatic Impairment Participants vs Part 2: Healthy Participants; Test type: Other; Ratio of Geometric LS Mean = 1.9375, 90% CI 2-sided [1.3919 to 2.6968] — Ratio of Geometric LS Mean for GSK2391220 (M2) (Mild hepatic impairment participants versus Healthy participants) has been presented
Statistical Analysis 3: Comparison: Part 2: Mild Hepatic Impairment Participants vs Part 2: Healthy Participants; Test type: Other; Ratio of Geometric LS Mean = 1.8312, 90% CI 2-sided [1.3342 to 2.5133] — Ratio of Geometric LS Mean for GSK2506104 (M3) (Mild hepatic impairment participants versus Healthy participants) has been presented
Statistical Analysis 4: Comparison: Part 2: Mild Hepatic Impairment Participants vs Part 2: Healthy Participants; Test type: Other; Ratio of Geometric LS Mean = 2.0030, 90% CI 2-sided [1.4654 to 2.7378] — Ratio of Geometric LS Mean for GSK2487818 (M4) (Mild hepatic impairment participants versus Healthy participants) has been presented
Statistical Analysis 5: Comparison: Part 2: Mild Hepatic Impairment Participants vs Part 2: Healthy Participants; Test type: Other; Ratio of Geometric LS Mean = 1.7113, 90% CI 2-sided [1.2818 to 2.2847] — Ratio of Geometric LS Mean for GSK2506102 (M5) (Mild hepatic impairment participants versus Healthy participants) has been presented
Statistical Analysis 6: Comparison: Part 2: Mild Hepatic Impairment Participants vs Part 2: Healthy Participants; Test type: Other; Ratio of Geometric LS Mean = 1.9740, 90% CI 2-sided [1.5365 to 2.5360] — Ratio of Geometric LS Mean for GSK2531398 (M6) (Mild hepatic impairment participants versus Healthy participants) has been presented
Statistical Analysis 7: Comparison: Part 2: Mild Hepatic Impairment Participants vs Part 2: Healthy Participants; Test type: Other; Ratio of Geometric LS Mean = 1.4603, 90% CI 2-sided [0.9081 to 2.3484] — Ratio of Geometric LS Mean for GSK2531401 (M13) (Mild hepatic impairment participants versus Healthy participants) has been presented

3. Primary Outcome: Part 1: Percentage of AUC (0-infinity) Obtained by Extrapolation (Percentage AUCex) of GSK1278863 and Its Metabolites
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK1278863 and its metabolites; GSK2391220 (M2), GSK2506104 (M3), GSK2487818 (M4), GSK2506102 (M5), GSK2531398 (M6), and GSK2531401 (M13). Pharmacokinetic parameters were determined using standard non-compartmental methods.
Time Frame: as for outcome 1
Population: Pharmacokinetic Population
Measure: Mean (Standard Deviation); unit: Percentage of AUCex
Arm/Group | Part 1: Moderate Hepatic Impairment Participants | Part 1: Healthy Participants
Number analyzed (Participants) | 8 | 8
Percentage of AUCex
  GSK1278863 | 0.0463 (0.03971) | 0.0486 (0.03445)
  GSK2391220 (M2) | 0.1919 (0.14164) | 0.4176 (0.38893)
  GSK2487818 (M4) | 0.5756 (0.89564) | 0.6763 (0.61031)
  GSK2506102 (M5) | 0.6147 (0.17403) | 2.1559 (2.01781)
  GSK2506104 (M3) | NA (NA) — Data was not calculable for the metabolite GSK2506104 (M3) due to matrix-related suppression during the bio-analysis of the Part 1 pharmacokinetic plasma samples. | NA (NA) — Data was not calculable for the metabolite GSK2506104 (M3) due to matrix-related suppression during the bio-analysis of the Part 1 pharmacokinetic plasma samples.
  GSK2531398 (M6) | 0.2598 (0.10004) | 0.3689 (0.26189)
  GSK2531401 (M13) | 0.2983 (0.27141) | 0.2787 (0.15617)

4. Primary Outcome: Part 2: Percentage AUCex of GSK1278863 and Its Metabolites
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK1278863 and its metabolites; GSK2391220 (M2), GSK2506104 (M3), GSK2487818 (M4), GSK2506102 (M5), GSK2531398 (M6), GSK2531401 (M13). Pharmacokinetic parameters were determined using standard non-compartmental methods.
Time Frame: as for outcome 1
Population: Pharmacokinetic Population. Only those participants with data available at specified time point were analyzed.
Measure: Mean (Standard Deviation); unit: Percentage of AUCex
Arm/Group | Part 2: Mild Hepatic Impairment Participants | Part 2: Healthy Participants
Number analyzed (Participants) | 8 | 7
Percentage of AUCex
  GSK1278863 | 0.1148 (0.26035) | 0.0601 (0.06032)
  GSK2391220 (M2) | 0.2943 (0.32698) | 0.8105 (1.60084)
  GSK2487818 (M4) | 0.2584 (0.30727) | 0.9054 (0.89147)
  GSK2506102 (M5) | 0.5138 (0.22859) | 1.5924 (1.69300)
  GSK2506104 (M3) | 0.2565 (0.28382) | 0.6875 (1.33005)
  GSK2531398 (M6) | 0.2915 (0.25350) | 0.9412 (0.94415)
  GSK2531401 (M13) | 0.2327 (0.23338) | 0.5256 (0.46352)

5. Primary Outcome: Part 1: Area Under the Concentration-time Curve From Time Zero (Pre-dose) to Last Time of Quantifiable Concentration (AUC [0-t]) of GSK1278863 and Its Metabolites
Description: as for outcome 4
Time Frame: as for outcome 1
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*nanogram per milliliter
Arm/Group | Part 1: Moderate Hepatic Impairment Participants | Part 1: Healthy Participants
Number analyzed (Participants) | 8 | 8
Hour*nanogram per milliliter
  GSK1278863 | 296.1035 (111.2) | 148.2504 (31.8)
  GSK2391220 (M2) | 77.4861 (57.0) | 46.9368 (31.0)
  GSK2487818 (M4) | 47.2803 (67.7) | 28.7930 (30.6)
  GSK2506102 (M5) | 16.7177 (43.9) | 11.0208 (30.9)
  GSK2506104 (M3) | NA (NA) — Data was not calculable for the metabolite GSK2506104 (M3) due to matrix-related suppression during the bio-analysis of the Part 1 pharmacokinetic plasma samples. | NA (NA) — Data was not calculable for the metabolite GSK2506104 (M3) due to matrix-related suppression during the bio-analysis of the Part 1 pharmacokinetic plasma samples.
  GSK2531398 (M6) | 33.8516 (49.3) | 20.8451 (27.8)
  GSK2531401 (M13) | 51.9052 (34.1) | 39.4939 (32.3)
Statistical Analysis 1: Comparison: Part 1: Moderate Hepatic Impairment Participants vs Part 1: Healthy Participants; Test type: Other; Ratio of Geometric LS Mean = 1.9973, 90% CI 2-sided [1.1061 to 3.6066] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Part 1: Moderate Hepatic Impairment Participants vs Part 1: Healthy Participants; Test type: Other; Ratio of Geometric LS Mean = 1.6509, 90% CI 2-sided [1.1285 to 2.4150] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Part 1: Moderate Hepatic Impairment Participants vs Part 1: Healthy Participants; Test type: Other; Ratio of Geometric LS Mean = 1.6421, 90% CI 2-sided [1.0732 to 2.5125] — [estimate comment as in outcome 1, analysis 3]
Statistical Analysis 4: Comparison: Part 1: Moderate Hepatic Impairment Participants vs Part 1: Healthy Participants; Test type: Other; Ratio of Geometric LS Mean = 1.5169, 90% CI 2-sided [1.0994 to 2.0930] — [estimate comment as in outcome 1, analysis 4]
Statistical Analysis 5: Comparison: Part 1: Moderate Hepatic Impairment Participants vs Part 1: Healthy Participants; Test type: Other; Ratio of Geometric LS Mean = 1.6240, 90% CI 2-sided [1.1599 to 2.2736] — [estimate comment as in outcome 1, analysis 5]
Statistical Analysis 6: Comparison: Part 1: Moderate Hepatic Impairment Participants vs Part 1: Healthy Participants; Test type: Other; Ratio of Geometric LS Mean = 1.3143, 90% CI 2-sided [0.9887 to 1.7470] — [estimate comment as in outcome 1, analysis 6]

6. Primary Outcome: Part 2: AUC (0-t) of GSK1278863 and Its Metabolites
Description: as for outcome 4
Time Frame: as for outcome 1
Population: Pharmacokinetic Population. Only those participants with data available at specified time point were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*nanogram per milliliter
Arm/Group | Part 2: Mild Hepatic Impairment Participants | Part 2: Healthy Participants
Number analyzed (Participants) | 8 | 7
Hour*nanogram per milliliter
  GSK1278863 | 299.5322 (39.9) | 205.6322 (37.2)
  GSK2391220 (M2) | 91.1105 (44.9) | 46.7771 (27.9)
  GSK2487818 (M4) | 63.4564 (40.3) | 31.4750 (29.0)
  GSK2506102 (M5) | 19.3023 (36.8) | 11.1555 (27.1)
  GSK2506104 (M3) | 91.5334 (41.2) | 49.7669 (29.2)
  GSK2531398 (M6) | 41.3456 (31.4) | 20.8080 (24.0)
  GSK2531401 (M13) | 46.5914 (66.8) | 31.8113 (41.3)
Statistical Analysis 1: Comparison: Part 2: Mild Hepatic Impairment Participants vs Part 2: Healthy Participants; Test type: Other; Ratio of Geometric LS Mean = 1.4566, 90% CI 2-sided [1.0344 to 2.0513] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Part 2: Mild Hepatic Impairment Participants vs Part 2: Healthy Participants; Test type: Other; Ratio of Geometric LS Mean = 1.9478, 90% CI 2-sided [1.3935 to 2.7224] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 3: Comparison: Part 2: Mild Hepatic Impairment Participants vs Part 2: Healthy Participants; Test type: Other; Ratio of Geometric LS Mean = 1.8392, 90% CI 2-sided [1.3350 to 2.5340] — [estimate comment as in outcome 2, analysis 3]
Statistical Analysis 4: Comparison: Part 2: Mild Hepatic Impairment Participants vs Part 2: Healthy Participants; Test type: Other; Ratio of Geometric LS Mean = 2.0161, 90% CI 2-sided [1.4711 to 2.7630] — [estimate comment as in outcome 2, analysis 4]
Statistical Analysis 5: Comparison: Part 2: Mild Hepatic Impairment Participants vs Part 2: Healthy Participants; Test type: Other; Ratio of Geometric LS Mean = 1.7303, 90% CI 2-sided [1.2932 to 2.3151] — [estimate comment as in outcome 2, analysis 5]
Statistical Analysis 6: Comparison: Part 2: Mild Hepatic Impairment Participants vs Part 2: Healthy Participants; Test type: Other; Ratio of Geometric LS Mean = 1.9870, 90% CI 2-sided [1.5426 to 2.5594] — [estimate comment as in outcome 2, analysis 6]
Statistical Analysis 7: Comparison: Part 2: Mild Hepatic Impairment Participants vs Part 2: Healthy Participants; Test type: Other; Ratio of Geometric LS Mean = 1.4646, 90% CI 2-sided [0.9086 to 2.3609] — [estimate comment as in outcome 2, analysis 7]

7. Primary Outcome: Part 1: Maximum Observed Concentration (Cmax) of GSK1278863 and Its Metabolites
Description: as for outcome 4
Time Frame: as for outcome 1
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Part 1: Moderate Hepatic Impairment Participants | Part 1: Healthy Participants
Number analyzed (Participants) | 8 | 8
Nanogram per milliliter
  GSK1278863 | 139.705 (108.8) | 70.607 (51.7)
  GSK2391220 (M2) | 13.046 (46.2) | 10.199 (28.7)
  GSK2487818 (M4) | 10.022 (55.0) | 8.025 (28.5)
  GSK2506102 (M5) | 2.650 (34.6) | 2.245 (23.0)
  GSK2506104 (M3) | NA (NA) — Data was not calculable for the metabolite GSK2506104 (M3) due to matrix-related suppression during the bio-analysis of the Part 1 pharmacokinetic plasma samples. | NA (NA) — Data was not calculable for the metabolite GSK2506104 (M3) due to matrix-related suppression during the bio-analysis of the Part 1 pharmacokinetic plasma samples.
  GSK2531398 (M6) | 5.946 (41.7) | 4.672 (24.1)
  GSK2531401 (M13) | 7.411 (35.0) | 7.120 (28.0)
Statistical Analysis 1: Comparison: Part 1: Moderate Hepatic Impairment Participants vs Part 1: Healthy Participants; Test type: Other; Ratio of Geometric LS Mean = 1.9786, 90% CI 2-sided [1.0557 to 3.7084] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Part 1: Moderate Hepatic Impairment Participants vs Part 1: Healthy Participants; Test type: Other; Ratio of Geometric LS Mean = 1.2791, 90% CI 2-sided [0.9241 to 1.7705] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Part 1: Moderate Hepatic Impairment Participants vs Part 1: Healthy Participants; Test type: Other; Ratio of Geometric LS Mean = 1.2487, 90% CI 2-sided [0.8675 to 1.7974] — [estimate comment as in outcome 1, analysis 3]
Statistical Analysis 4: Comparison: Part 1: Moderate Hepatic Impairment Participants vs Part 1: Healthy Participants; Test type: Other; Ratio of Geometric LS Mean = 1.1802, 90% CI 2-sided [0.9165 to 1.5197] — [estimate comment as in outcome 1, analysis 4]
Statistical Analysis 5: Comparison: Part 1: Moderate Hepatic Impairment Participants vs Part 1: Healthy Participants; Test type: Other; Ratio of Geometric LS Mean = 1.2726, 90% CI 2-sided [0.9520 to 1.7012] — [estimate comment as in outcome 1, analysis 5]
Statistical Analysis 6: Comparison: Part 1: Moderate Hepatic Impairment Participants vs Part 1: Healthy Participants; Test type: Other; Ratio of Geometric LS Mean = 1.0409, 90% CI 2-sided [0.7927 to 1.3668] — [estimate comment as in outcome 1, analysis 6]

8. Primary Outcome: Part 2: Cmax of GSK1278863 and Its Metabolites.
Description: as for outcome 3
Time Frame: as for outcome 1
Population: Pharmacokinetic Population. Only those participants with data available at specified time point were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Part 2: Mild Hepatic Impairment Participants | Part 2: Healthy Participants
Number analyzed (Participants) | 8 | 7
Nanogram per milliliter
  GSK1278863 | 113.232 (42.6) | 112.142 (35.7)
  GSK2391220 (M2) | 15.792 (40.8) | 8.846 (40.0)
  GSK2487818 (M4) | 13.614 (34.7) | 7.723 (35.6)
  GSK2506102 (M5) | 3.241 (35.7) | 1.975 (33.4)
  GSK2506104 (M3) | 15.475 (38.8) | 8.926 (37.9)
  GSK2531398 (M6) | 7.333 (28.2) | 4.010 (31.7)
  GSK2531401 (M13) | 6.791 (65.5) | 5.081 (43.4)
Statistical Analysis 1: Comparison: Part 2: Mild Hepatic Impairment Participants vs Part 2: Healthy Participants; Test type: Other; Ratio of Geometric LS Mean = 1.0097, 90% CI 2-sided [0.7122 to 1.4316] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Part 2: Mild Hepatic Impairment Participants vs Part 2: Healthy Participants; Test type: Other; Ratio of Geometric LS Mean = 1.7852, 90% CI 2-sided [1.2498 to 2.5498] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 3: Comparison: Part 2: Mild Hepatic Impairment Participants vs Part 2: Healthy Participants; Test type: Other; Ratio of Geometric LS Mean = 1.7337, 90% CI 2-sided [1.2343 to 2.4353] — [estimate comment as in outcome 2, analysis 3]
Statistical Analysis 4: Comparison: Part 2: Mild Hepatic Impairment Participants vs Part 2: Healthy Participants; Test type: Other; Ratio of Geometric LS Mean = 1.7628, 90% CI 2-sided [1.2898 to 2.4092] — [estimate comment as in outcome 2, analysis 4]
Statistical Analysis 5: Comparison: Part 2: Mild Hepatic Impairment Participants vs Part 2: Healthy Participants; Test type: Other; Ratio of Geometric LS Mean = 1.6413, 90% CI 2-sided [1.2055 to 2.2347] — [estimate comment as in outcome 2, analysis 5]
Statistical Analysis 6: Comparison: Part 2: Mild Hepatic Impairment Participants vs Part 2: Healthy Participants; Test type: Other; Ratio of Geometric LS Mean = 1.8289, 90% CI 2-sided [1.3992 to 2.3904] — [estimate comment as in outcome 2, analysis 6]
Statistical Analysis 7: Comparison: Part 2: Mild Hepatic Impairment Participants vs Part 2: Healthy Participants; Test type: Other; Ratio of Geometric LS Mean = 1.3367, 90% CI 2-sided [0.8288 to 2.1557] — [estimate comment as in outcome 2, analysis 7]

9. Primary Outcome: Part 1: Apparent Terminal Phase Half-life (t1/2) of GSK1278863 and Its Metabolites
Description: as for outcome 4
Time Frame: as for outcome 1
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Part 1: Moderate Hepatic Impairment Participants | Part 1: Healthy Participants
Number analyzed (Participants) | 8 | 8
Hours
  GSK1278863 | 3.9867 (33.2) | 4.4054 (29.8)
  GSK2391220 (M2) | 4.1830 (26.9) | 5.6415 (37.1)
  GSK2487818 (M4) | 2.6559 (38.3) | 3.6385 (83.8)
  GSK2506102 (M5) | 3.1966 (23.4) | 2.7314 (36.4)
  GSK2506104 (M3) | NA (NA) — Data was not calculable for the metabolite GSK2506104 (M3) due to matrix-related suppression during the bio-analysis of the Part 1 pharmacokinetic plasma samples. | NA (NA) — Data was not calculable for the metabolite GSK2506104 (M3) due to matrix-related suppression during the bio-analysis of the Part 1 pharmacokinetic plasma samples.
  GSK2531398 (M6) | 3.1287 (26.0) | 3.2641 (56.3)
  GSK2531401 (M13) | 3.9432 (22.8) | 3.9414 (33.1)
Statistical Analysis 1: Comparison: Part 1: Moderate Hepatic Impairment Participants vs Part 1: Healthy Participants; Test type: Other; Ratio of Geometric LS Mean = 0.9050, 90% CI 2-sided [0.6900 to 1.1869] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Part 1: Moderate Hepatic Impairment Participants vs Part 1: Healthy Participants; Test type: Other; Ratio of Geometric LS Mean = 0.7415, 90% CI 2-sided [0.5617 to 0.9787] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Part 1: Moderate Hepatic Impairment Participants vs Part 1: Healthy Participants; Test type: Other; Ratio of Geometric LS Mean = 0.7299, 90% CI 2-sided [0.4387 to 1.2145] — [estimate comment as in outcome 1, analysis 3]
Statistical Analysis 4: Comparison: Part 1: Moderate Hepatic Impairment Participants vs Part 1: Healthy Participants; Test type: Other; Ratio of Geometric LS Mean = 1.1703, 90% CI 2-sided [0.9000 to 1.5219] — [estimate comment as in outcome 1, analysis 4]
Statistical Analysis 5: Comparison: Part 1: Moderate Hepatic Impairment Participants vs Part 1: Healthy Participants; Test type: Other; Ratio of Geometric LS Mean = 0.9585, 90% CI 2-sided [0.6664 to 1.3786] — [estimate comment as in outcome 1, analysis 5]
Statistical Analysis 6: Comparison: Part 1: Moderate Hepatic Impairment Participants vs Part 1: Healthy Participants; Test type: Other; Ratio of Geometric LS Mean = 1.0004, 90% CI 2-sided [0.7833 to 1.2778] — [estimate comment as in outcome 1, analysis 6]

10. Primary Outcome: Part 2: T1/2 of GSK1278863 and Its Metabolites
Description: as for outcome 4
Time Frame: as for outcome 1
Population: Pharmacokinetic Population. Only those participants with data available at specified time point were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Part 2: Mild Hepatic Impairment Participants | Part 2: Healthy Participants
Number analyzed (Participants) | 8 | 7
Hours
  GSK1278863 | 4.5251 (27.4) | 4.2792 (38.7)
  GSK2391220 (M2) | 4.8118 (21.2) | 4.7439 (49.6)
  GSK2487818 (M4) | 4.1059 (47.8) | 3.0578 (88.9)
  GSK2506102 (M5) | 3.4087 (30.8) | 3.3108 (56.7)
  GSK2506104 (M3) | 4.6675 (20.2) | 4.4967 (45.0)
  GSK2531398 (M6) | 3.8096 (38.4) | 2.9947 (57.1)
  GSK2531401 (M13) | 4.2869 (21.2) | 3.5510 (34.2)
Statistical Analysis 1: Comparison: Part 2: Mild Hepatic Impairment Participants vs Part 2: Healthy Participants; Test type: Other; Ratio of Geometric LS Mean = 1.0574, 90% CI 2-sided [0.7876 to 1.4197] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Part 2: Mild Hepatic Impairment Participants vs Part 2: Healthy Participants; Test type: Other; Ratio of Geometric LS Mean = 1.0143, 90% CI 2-sided [0.7332 to 1.4032] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 3: Comparison: Part 2: Mild Hepatic Impairment Participants vs Part 2: Healthy Participants; Test type: Other; Ratio of Geometric LS Mean = 1.0380, 90% CI 2-sided [0.7695 to 1.4002] — [estimate comment as in outcome 2, analysis 3]
Statistical Analysis 4: Comparison: Part 2: Mild Hepatic Impairment Participants vs Part 2: Healthy Participants; Test type: Other; Ratio of Geometric LS Mean = 1.3427, 90% CI 2-sided [0.7635 to 2.3615] — [estimate comment as in outcome 2, analysis 4]
Statistical Analysis 5: Comparison: Part 2: Mild Hepatic Impairment Participants vs Part 2: Healthy Participants; Test type: Other; Ratio of Geometric LS Mean = 1.0296, 90% CI 2-sided [0.6996 to 1.5151] — [estimate comment as in outcome 2, analysis 5]
Statistical Analysis 6: Comparison: Part 2: Mild Hepatic Impairment Participants vs Part 2: Healthy Participants; Test type: Other; Ratio of Geometric LS Mean = 1.2721, 90% CI 2-sided [0.8409 to 1.9245] — [estimate comment as in outcome 2, analysis 6]
Statistical Analysis 7: Comparison: Part 2: Mild Hepatic Impairment Participants vs Part 2: Healthy Participants; Test type: Other; Ratio of Geometric LS Mean = 1.2072, 90% CI 2-sided [0.9398 to 1.5508] — [estimate comment as in outcome 2, analysis 7]

11. Primary Outcome: Part 1: Time of Occurrence of Cmax (Tmax) of GSK1278863 and Its Metabolites
Description: as for outcome 4
Time Frame: as for outcome 1
Population: Pharmacokinetic Population
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 1: Moderate Hepatic Impairment Participants | Part 1: Healthy Participants
Number analyzed (Participants) | 8 | 8
Hours
  GSK1278863 | 1.50 [1.0 to 3.0] | 2.00 [1.0 to 3.0]
  GSK2391220 (M2) | 3.00 [3.0 to 6.0] | 3.50 [2.0 to 4.0]
  GSK2487818 (M4) | 3.00 [2.0 to 6.0] | 3.00 [1.5 to 4.0]
  GSK2506102 (M5) | 3.50 [3.0 to 6.0] | 4.00 [2.0 to 4.0]
  GSK2506104 (M3) | NA [NA to NA] — Data was not calculable for the metabolite GSK2506104 (M3) due to matrix-related suppression during the bio-analysis of the Part 1 pharmacokinetic plasma samples. | NA [NA to NA] — Data was not calculable for the metabolite GSK2506104 (M3) due to matrix-related suppression during the bio-analysis of the Part 1 pharmacokinetic plasma samples.
  GSK2531398 (M6) | 3.50 [3.0 to 6.0] | 3.50 [2.0 to 4.0]
  GSK2531401 (M13) | 4.00 [3.0 to 6.0] | 4.00 [3.0 to 6.0]
Statistical Analysis 1: Comparison: Part 1: Moderate Hepatic Impairment Participants vs Part 1: Healthy Participants; Test type: Other; p = 0.6822, Wilcoxon (Mann-Whitney) — P-value was based on Mann-Whitney U test (exact Wilcoxon rank sum test); Median Difference (Final Values) = 0.00, 90% CI 2-sided [-1.00 to 0.50] — Median Difference in GSK1278863 (Moderate hepatic impairment participants versus Healthy participants) has been presented
Statistical Analysis 2: Comparison: Part 1: Moderate Hepatic Impairment Participants vs Part 1: Healthy Participants; Test type: Other; p = 0.5767, Wilcoxon (Mann-Whitney) — P-value was based on Mann-Whitney U test (exact Wilcoxon rank sum test); Median Difference (Final Values) = 0.00, 90% CI 2-sided [-1.00 to 1.00] — Median Difference in GSK2391220 (M2)(Moderate hepatic impairment participants versus Healthy participants) has been presented
Statistical Analysis 3: Comparison: Part 1: Moderate Hepatic Impairment Participants vs Part 1: Healthy Participants; Test type: Other; p = 0.5880, Wilcoxon (Mann-Whitney) — P-value was based on Mann-Whitney U test (exact Wilcoxon rank sum test); Median Difference (Final Values) = 0.00, 90% CI 2-sided [-1.00 to 1.50] — Median Difference in GSK2487818 (M4)(Moderate hepatic impairment participants versus Healthy participants) has been presented
Statistical Analysis 4: Comparison: Part 1: Moderate Hepatic Impairment Participants vs Part 1: Healthy Participants; Test type: Other; p = 0.7716, Wilcoxon (Mann-Whitney) — P-value was based on Mann-Whitney U test (exact Wilcoxon rank sum test); Median Difference (Final Values) = 0.00, 90% CI 2-sided [-1.00 to 1.00] — Median Difference in GSK2506102 (M5)(Moderate hepatic impairment participants versus Healthy participants) has been presented
Statistical Analysis 5: Comparison: Part 1: Moderate Hepatic Impairment Participants vs Part 1: Healthy Participants; Test type: Other; p = 0.4093, Wilcoxon (Mann-Whitney) — P-value was based on Mann-Whitney U test (exact Wilcoxon rank sum test); Median Difference (Final Values) = 0.50, 90% CI 2-sided [-1.00 to 2.00] — Median Difference in GSK2531398 (M6) (Moderate hepatic impairment participants versus Healthy participants) has been presented
Statistical Analysis 6: Comparison: Part 1: Moderate Hepatic Impairment Participants vs Part 1: Healthy Participants; Test type: Other; p = 0.9837, Wilcoxon (Mann-Whitney) — P-value was based on Mann-Whitney U test (exact Wilcoxon rank sum test); Median Difference (Final Values) = 0.00, 90% CI 2-sided [-1.00 to 1.00] — Median Difference in GSK2531401 (M13) (Moderate hepatic impairment participants versus Healthy participants) has been presented

12. Primary Outcome: Part 2: Tmax of GSK1278863 and Its Metabolites
Description: as for outcome 4
Time Frame: as for outcome 1
Population: Pharmacokinetic Population. Only those participants with data available at specified time point were analyzed.
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 2: Mild Hepatic Impairment Participants | Part 2: Healthy Participants
Number analyzed (Participants) | 8 | 7
Hours
  GSK1278863 | 1.50 [1.0 to 3.0] | 1.50 [1.0 to 4.0]
  GSK2391220 (M2) | 3.00 [3.0 to 4.0] | 3.00 [2.0 to 4.0]
  GSK2487818 (M4) | 3.00 [2.0 to 4.0] | 3.00 [2.0 to 4.0]
  GSK2506102 (M5) | 3.50 [3.0 to 4.0] | 3.00 [2.0 to 6.0]
  GSK2506104 (M3) | 3.50 [3.0 to 4.0] | 3.00 [2.0 to 6.0]
  GSK2531398 (M6) | 3.00 [3.0 to 4.0] | 3.00 [2.0 to 6.0]
  GSK2531401 (M13) | 4.00 [3.0 to 4.0] | 4.00 [3.0 to 6.0]
Statistical Analysis 1: Comparison: Part 2: Mild Hepatic Impairment Participants vs Part 2: Healthy Participants; Test type: Other; p = 0.6224, Wilcoxon (Mann-Whitney) — P-value was based on Mann-Whitney U test (exact Wilcoxon rank sum test); Median Difference (Final Values) = 0.00, 90% CI 2-sided [-1.00 to 0.50] — Median Difference in GSK1278863 (Mild hepatic impairment participants versus Healthy participants) has been presented
Statistical Analysis 2: Comparison: Part 2: Mild Hepatic Impairment Participants vs Part 2: Healthy Participants; Test type: Other; p = 0.8042, Wilcoxon (Mann-Whitney) — P-value was based on Mann-Whitney U test (exact Wilcoxon rank sum test); Median Difference (Final Values) = 0.00, 90% CI 2-sided [-1.00 to 0.00] — Median Difference in GSK2391220 (M2) (Mild hepatic impairment participants versus Healthy participants) has been presented
Statistical Analysis 3: Comparison: Part 2: Mild Hepatic Impairment Participants vs Part 2: Healthy Participants; Test type: Other; p = 0.8423, Wilcoxon (Mann-Whitney) — P-value was based on Mann-Whitney U test (exact Wilcoxon rank sum test); Median Difference (Final Values) = 0.00, 90% CI 2-sided [-1.00 to 1.00] — Median Difference in GSK2506104 (M3) (Mild hepatic impairment participants versus Healthy participants) has been presented
Statistical Analysis 4: Comparison: Part 2: Mild Hepatic Impairment Participants vs Part 2: Healthy Participants; Test type: Other; p = 0.5207, Wilcoxon (Mann-Whitney) — P-value was based on Mann-Whitney U test (exact Wilcoxon rank sum test); Median Difference (Final Values) = 0.00, 90% CI 2-sided [-1.00 to 1.00] — Median Difference in GSK2487818 (M4) (Mild hepatic impairment participants versus Healthy participants) has been presented
Statistical Analysis 5: Comparison: Part 2: Mild Hepatic Impairment Participants vs Part 2: Healthy Participants; Test type: Other; p = 0.8423, Wilcoxon (Mann-Whitney) — P-value was based on Mann-Whitney U test (exact Wilcoxon rank sum test); Median Difference (Final Values) = 0.00, 90% CI 2-sided [-1.00 to 1.00] — Median Difference in GSK2506102 (M5) (Mild hepatic impairment participants versus Healthy participants) has been presented
Statistical Analysis 6: Comparison: Part 2: Mild Hepatic Impairment Participants vs Part 2: Healthy Participants; Test type: Other; p = 1.0000, Wilcoxon (Mann-Whitney) — P-value was based on Mann-Whitney U test (exact Wilcoxon rank sum test); Median Difference (Final Values) = 0.00, 90% CI 2-sided [-1.00 to 1.00] — Median Difference in GSK2531398 (M6) (Mild hepatic impairment participants versus Healthy participants) has been presented
Statistical Analysis 7: Comparison: Part 2: Mild Hepatic Impairment Participants vs Part 2: Healthy Participants; Test type: Other; p = 0.8042, Wilcoxon (Mann-Whitney) — P-value was based on Mann-Whitney U test (exact Wilcoxon rank sum test); Median Difference (Final Values) = 0.00, 90% CI 2-sided [0.00 to 1.00] — Median Difference in GSK2531401 (M13) (Mild hepatic impairment participants versus Healthy participants) has been presented

13. Primary Outcome: Part 1: Unbound Concentration in Plasma of GSK1278863 and Its Metabolites
Description: as for outcome 4
Time Frame: 3 hours, 12 hours and 24 hours post-dose
Population: Pharmacokinetic Population
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter
Arm/Group | Part 1: Moderate Hepatic Impairment Participants | Part 1: Healthy Participants
Number analyzed (Participants) | 8 | 8
Nanograms per milliliter
  GSK1278863; 3 hours | 0.27989 (0.261668) | 0.11076 (0.070114)
  GSK1278863; 12 hours | NA (NA) — Mean and Standard Deviation were not calculable because concentration values were below detectable levels, but were imputed in the analysis. | NA (NA) — Mean and Standard Deviation were not calculable because concentration values were below detectable levels, but were imputed in the analysis.
  GSK1278863; 24 hours | NA (NA) — Mean and Standard Deviation were not calculable because concentration values were below detectable levels, but were imputed in the analysis. | NA (NA) — Mean and Standard Deviation were not calculable because concentration values were below detectable levels, but were imputed in the analysis.
  GSK2391220 (M2); 3 hours | 4.47750 (1.779468) | 2.85875 (1.129961)
  GSK2391220 (M2); 12 hours | 0.76525 (0.656087) | 0.22463 (0.119826)
  GSK2391220 (M2); 24 hours | 0.06460 (0.089209) | 0.00963 (0.017963)
  GSK2487818 (M4); 3 hours | 3.24463 (1.506964) | 1.86813 (0.760479)
  GSK2487818 (M4); 12 hours | 0.29301 (0.338773) | 0.04769 (0.031411)
  GSK2487818 (M4); 24 hours | 0.01201 (0.023617) | NA (NA) — Mean and Standard Deviation were not calculable because concentration values were below detectable levels, but were imputed in the analysis.
  GSK2506102 (M5); 3 hours | 0.64588 (0.242321) | 0.43175 (0.165059)
  GSK2506102 (M5); 12 hours | 0.13024 (0.109089) | 0.04143 (0.031140)
  GSK2506102 (M5); 24 hours | 0.00923 (0.026092) | NA (NA) — Mean and Standard Deviation were not calculable because concentration values were below detectable levels, but were imputed in the analysis.
  GSK2506104 (M3); 3 hours | 3.86250 (1.402241) | 2.57000 (1.010262)
  GSK2506104 (M3); 12 hours | 0.71075 (0.601452) | 0.23938 (0.121781)
  GSK2506104 (M3); 24 hours | 0.06315 (0.104994) | 0.00829 (0.015374)
  GSK2531398 (M6); 3 hours | 1.42725 (0.552287) | 0.89338 (0.334179)
  GSK2531398 (M6); 12 hours | 0.22973 (0.199514) | 0.06548 (0.035504)
  GSK2531398 (M6); 24 hours | 0.01470 (0.028580) | NA (NA) — Mean and Standard Deviation were not calculable because concentration values were below detectable levels, but were imputed in the analysis.
  GSK2531401 (M13); 3 hours | 2.25375 (0.646771) | 2.03738 (0.807331)
  GSK2531401 (M13); 12 hours | 0.63125 (0.379804) | 0.32075 (0.163981)
  GSK2531401 (M13); 24 hours | 0.07580 (0.110738) | 0.01053 (0.020023)

14. Primary Outcome: Part 2: Unbound Concentration in Plasma of GSK1278863 and Its Metabolites
Description: as for outcome 4
Time Frame: 3 hours, 12 hours and 24 hours post-dose
Population: Pharmacokinetic Population. Only those participants with data available at specified time point were analyzed (represented by n=X in category titles).
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter
Arm/Group | Part 2: Mild Hepatic Impairment Participants | Part 2: Healthy Participants
Number analyzed (Participants) | 8 | 8
Nanograms per milliliter
  GSK1278863; 3 hours; n=6, 6: number analyzed (Participants) | 6 | 6
  GSK1278863; 3 hours; n=6, 6 | 1.24213 (2.475347) | 0.15692 (0.138726)
  GSK1278863; 12 hours; n=7, 6: number analyzed (Participants) | 7 | 6
  GSK1278863; 12 hours; n=7, 6 | 0.04343 (0.114901) | 0.01527 (0.037396)
  GSK1278863; 24 hours; n=7, 6: number analyzed (Participants) | 7 | 6
  GSK1278863; 24 hours; n=7, 6 | NA (NA) — Mean and Standard Deviation were not calculable because concentration values were below detectable levels, but were imputed in the analysis. | NA (NA) — Mean and Standard Deviation were not calculable because concentration values were below detectable levels, but were imputed in the analysis.
  GSK2391220 (M2); 3 hours; n=8, 7: number analyzed (Participants) | 8 | 7
  GSK2391220 (M2); 3 hours; n=8, 7 | 5.32625 (2.139472) | 2.13700 (1.276959)
  GSK2391220 (M2); 12 hours; n=8, 7: number analyzed (Participants) | 8 | 7
  GSK2391220 (M2); 12 hours; n=8, 7 | 0.81263 (0.600031) | 0.24371 (0.079803)
  GSK2391220 (M2); 24 hours; n=8, 7: number analyzed (Participants) | 8 | 7
  GSK2391220 (M2); 24 hours; n=8, 7 | 0.30654 (0.729605) | NA (NA) — Mean and Standard Deviation were not calculable because concentration values were below detectable levels, but were imputed in the analysis.
  GSK2487818 (M4); 3 hours; n=8,7: number analyzed (Participants) | 8 | 7
  GSK2487818 (M4); 3 hours; n=8,7 | 3.91375 (1.441219) | 1.57633 (0.937244)
  GSK2487818 (M4); 12 hours; n=8,7: number analyzed (Participants) | 8 | 7
  GSK2487818 (M4); 12 hours; n=8,7 | 0.40141 (0.560638) | 0.07793 (0.033300)
  GSK2487818 (M4); 24 hours; n=8,7: number analyzed (Participants) | 8 | 7
  GSK2487818 (M4); 24 hours; n=8,7 | 0.00839 (0.015586) | 0.00454 (0.012019)
  GSK2506102 (M5); 3 hours; n=8,7: number analyzed (Participants) | 8 | 7
  GSK2506102 (M5); 3 hours; n=8,7 | 0.78213 (0.314177) | 0.31091 (0.213793)
  GSK2506102 (M5); 12 hours; n=8,7: number analyzed (Participants) | 8 | 7
  GSK2506102 (M5); 12 hours; n=8,7 | 0.25856 (0.425759) | 0.04796 (0.035510)
  GSK2506102 (M5); 24 hours; n=8,7: number analyzed (Participants) | 8 | 7
  GSK2506102 (M5); 24 hours; n=8,7 | NA (NA) — Mean and Standard Deviation were not calculable because concentration values were below detectable levels, but were imputed in the analysis. | NA (NA) — Mean and Standard Deviation were not calculable because concentration values were below detectable levels, but were imputed in the analysis.
  GSK2506104 (M3); 3 hours; n=8,7: number analyzed (Participants) | 8 | 7
  GSK2506104 (M3); 3 hours; n=8,7 | 4.68625 (1.839883) | 1.94271 (1.262970)
  GSK2506104 (M3); 12 hours; n=8,7: number analyzed (Participants) | 8 | 7
  GSK2506104 (M3); 12 hours; n=8,7 | 0.75350 (0.496638) | 0.27014 (0.122830)
  GSK2506104 (M3); 24 hours; n=8,7: number analyzed (Participants) | 8 | 7
  GSK2506104 (M3); 24 hours; n=8,7 | 0.04093 (0.029445) | 0.00819 (0.021657)
  GSK2531398 (M6); 3 hours; n=8,7: number analyzed (Participants) | 8 | 7
  GSK2531398 (M6); 3 hours; n=8,7 | 1.86763 (0.713958) | 0.73530 (0.451869)
  GSK2531398 (M6); 12 hours; n=8,7: number analyzed (Participants) | 8 | 7
  GSK2531398 (M6); 12 hours; n=8,7 | 0.34200 (0.412505) | 0.07879 (0.023474)
  GSK2531398 (M6); 24 hours; n=8,7: number analyzed (Participants) | 8 | 7
  GSK2531398 (M6); 24 hours; n=8,7 | NA (NA) — Mean and Standard Deviation were not calculable because concentration values were below detectable levels, but were imputed in the analysis. | NA (NA) — Mean and Standard Deviation were not calculable because concentration values were below detectable levels, but were imputed in the analysis.
  GSK2531401 (M13); 3 hours; n=8,7: number analyzed (Participants) | 8 | 7
  GSK2531401 (M13); 3 hours; n=8,7 | 2.47825 (0.965944) | 1.26771 (0.871839)
  GSK2531401 (M13); 12 hours; n=8,7: number analyzed (Participants) | 8 | 7
  GSK2531401 (M13); 12 hours; n=8,7 | 0.75363 (0.597207) | 0.29429 (0.153615)
  GSK2531401 (M13); 24 hours; n=8,7: number analyzed (Participants) | 8 | 7
  GSK2531401 (M13); 24 hours; n=8,7 | 0.29830 (0.720919) | 0.00454 (0.012019)

15. Primary Outcome: Part 1: Unbound Fraction in Plasma of GSK1278863 and Its Metabolites
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK1278863 and its metabolites; GSK2391220 (M2), GSK2506104 (M3), GSK2487818, GSK2506102, GSK2531398 (M6), GSK2531401 (M13). Pharmacokinetic parameters were determined using standard non-compartmental methods. Unbound fraction is the percentage of unbound drug in plasma calculated as unbound concentration divided by total concentration.
Time Frame: 3 hours, 12 hours and 24 hours post-dose
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: Percentage of unbound drug in plasma
Arm/Group | Part 1: Moderate Hepatic Impairment Participants | Part 1: Healthy Participants
Number analyzed (Participants) | 8 | 8
Percentage of unbound drug in plasma
  GSK1278863; 3 hours; n=8, 8 | 0.0034 (0.00109) | 0.0028 (0.00019)
  GSK1278863; 12 hours; n=8, 8 | NA (NA) — Mean and Standard Deviation were not calculable because concentration values were below detectable levels, but were imputed in the analysis. | NA (NA) — Mean and Standard Deviation were not calculable because concentration values were below detectable levels, but were imputed in the analysis.
  GSK1278863; 24 hours; n=8,8 | NA (NA) — Mean and Standard Deviation were not calculable because concentration values were below detectable levels, but were imputed in the analysis. | NA (NA) — Mean and Standard Deviation were not calculable because concentration values were below detectable levels, but were imputed in the analysis.
  GSK2391220 (M2); 3 hours; n=8,8 | 0.3379 (0.03573) | 0.3495 (0.05135)
  GSK2391220 (M2); 12 hours; n=8,8 | 0.3540 (0.02186) | 0.3355 (0.02172)
  GSK2391220 (M2); 24 hours; n=4,2: number analyzed (Participants) | 4 | 2
  GSK2391220 (M2); 24 hours; n=4,2 | 0.3861 (0.02827) | 0.3902 (0.07149)
  GSK2487818 (M4); 3 hours; n=8,8 | 0.3080 (0.03085) | 0.2925 (0.01981)
  GSK2487818 (M4); 12 hours; n=8,7: number analyzed (Participants) | 8 | 7
  GSK2487818 (M4); 12 hours; n=8,7 | 0.3071 (0.03419) | 0.2402 (0.02431)
  GSK2487818 (M4); 24 hours; n=2,8: number analyzed (Participants) | 2 | 8
  GSK2487818 (M4); 24 hours; n=2,8 | 0.3508 (0.00191) | NA (NA) — Mean and Standard Deviation were not calculable because concentration values were below detectable levels, but were imputed in the analysis.
  GSK2506102 (M5); 3 hours; n=8, 8 | 0.2565 (0.04573) | 0.2441 (0.03397)
  GSK2506102 (M5); 12 hours; n=8, 6: number analyzed (Participants) | 8 | 6
  GSK2506102 (M5); 12 hours; n=8, 6 | 0.2517 (0.04022) | 0.2335 (0.02679)
  GSK2506102 (M5); 24 hours; n=1, 8: number analyzed (Participants) | 1 | 8
  GSK2506102 (M5); 24 hours; n=1, 8 | 0.2723 (NA) — Data was not available as standard deviation could not be calculated for single participant. | NA (NA) — Mean and Standard Deviation were not calculable because concentration values were below detectable levels, but were imputed in the analysis.
  GSK2506104 (M3); 3 hours; n=8, 8 | NA (NA) — Mean and Standard Deviation were not calculable because concentration values were below detectable levels, but were imputed in the analysis. | NA (NA) — Mean and Standard Deviation were not calculable because concentration values were below detectable levels, but were imputed in the analysis.
  GSK2506104 (M3); 12 hours; n=8, 8 | NA (NA) — Mean and Standard Deviation were not calculable because concentration values were below detectable levels, but were imputed in the analysis. | NA (NA) — Mean and Standard Deviation were not calculable because concentration values were below detectable levels, but were imputed in the analysis.
  GSK2506104 (M3); 24 hours; n=8, 8 | NA (NA) — Mean and Standard Deviation were not calculable because concentration values were below detectable levels, but were imputed in the analysis. | NA (NA) — Mean and Standard Deviation were not calculable because concentration values were below detectable levels, but were imputed in the analysis.
  GSK2531398 (M6); 3 hours; n=8, 8 | 0.2469 (0.04315) | 0.2461 (0.03264)
  GSK2531398 (M6); 12 hours; n=8, 8 | 0.2550 (0.03166) | 0.2295 (0.01509)
  GSK2531398 (M6); 24 hours; n=2, 8: number analyzed (Participants) | 2 | 8
  GSK2531398 (M6); 24 hours; n=2, 8 | 0.3005 (0.03734) | NA (NA) — Mean and Standard Deviation were not calculable because concentration values were below detectable levels, but were imputed in the analysis.
  GSK2531401 (M13); 3 hours; n=8, 8 | 0.3519 (0.04431) | 0.3844 (0.06838)
  GSK2531401 (M13); 12 hours; n=8, 8 | 0.3771 (0.02114) | 0.3565 (0.02558)
  GSK2531401 (M13); 24 hours; n=6, 2: number analyzed (Participants) | 6 | 2
  GSK2531401 (M13); 24 hours; n=6, 2 | 0.3817 (0.04449) | 0.3716 (0.02411)

16. Primary Outcome: Part 2: Unbound Fraction in Plasma of GSK1278863 and Its Metabolites
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK1278863 and its metabolites (GSK2391220 (M2), GSK2506104 (M3), GSK2487818 (M4), GSK2506102 (M5), GSK2531398 (M6), GSK2531401 (M13)). Pharmacokinetic parameters were determined using standard non-compartmental methods. Unbound fraction is the percentage of unbound drug in plasma calculated as unbound concentration divided by total concentration.
Time Frame: 3 hours, 12 hours and 24 hours post-dose
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: Percentage of unbound drug in plasma
Arm/Group | Part 2: Mild Hepatic Impairment Participants | Part 2: Healthy Participants
Number analyzed (Participants) | 8 | 8
Percentage of unbound drug in plasma
  GSK1278863; 3 hours; n=6, 6: number analyzed (Participants) | 6 | 6
  GSK1278863; 3 hours; n=6, 6 | 0.0134 (0.02369) | 0.0032 (0.00090)
  GSK1278863; 12 hours; n=1, 1: number analyzed (Participants) | 1 | 1
  GSK1278863; 12 hours; n=1, 1 | 0.1231 (NA) — Data was not available as standard deviation could not be calculated for single participant.. | 0.1246 (NA) — Data was not available as standard deviation could not be calculated for single participant..
  GSK1278863; 24 hours; n=8,7: number analyzed (Participants) | 8 | 7
  GSK1278863; 24 hours; n=8,7 | NA (NA) — Mean and Standard Deviation were not calculable because concentration values were below detectable levels, but were imputed in the analysis. | NA (NA) — Mean and Standard Deviation were not calculable because concentration values were below detectable levels, but were imputed in the analysis.
  GSK2391220 (M2); 3 hours; n=8, 7: number analyzed (Participants) | 8 | 7
  GSK2391220 (M2); 3 hours; n=8, 7 | 0.3191 (0.02263) | 0.3343 (0.06101)
  GSK2391220 (M2); 12 hours; n=7, 7: number analyzed (Participants) | 7 | 7
  GSK2391220 (M2); 12 hours; n=7, 7 | 0.3305 (0.03497) | 0.3174 (0.02174)
  GSK2391220 (M2); 24 hours; n=5, 7: number analyzed (Participants) | 5 | 7
  GSK2391220 (M2); 24 hours; n=5, 7 | 0.4099 (0.04797) | NA (NA) — Mean and Standard Deviation were not calculable because concentration values were below detectable levels, but were imputed in the analysis.
  GSK2487818 (M4); 3 hours; n=8, 7: number analyzed (Participants) | 8 | 7
  GSK2487818 (M4); 3 hours; n=8, 7 | 0.2762 (0.02792) | 0.2857 (0.03897)
  GSK2487818 (M4); 12 hours; n=7, 7: number analyzed (Participants) | 7 | 7
  GSK2487818 (M4); 12 hours; n=7, 7 | 0.2850 (0.03110) | 0.2766 (0.03608)
  GSK2487818 (M4); 24 hours; n=2, 1: number analyzed (Participants) | 2 | 1
  GSK2487818 (M4); 24 hours; n=2, 1 | 0.3116 (0.07106) | 0.3387 (NA) — Data was not available as standard deviation could not be calculated for single participant.
  GSK2506102 (M5); 3 hours; n=8, 6: number analyzed (Participants) | 8 | 6
  GSK2506102 (M5); 3 hours; n=8, 6 | 0.2339 (0.02704) | 0.2171 (0.06728)
  GSK2506102 (M5); 12 hours; n=7, 6: number analyzed (Participants) | 7 | 6
  GSK2506102 (M5); 12 hours; n=7, 6 | 0.2483 (0.03166) | 0.2191 (0.02903)
  GSK2506102 (M5); 24 hours; n=8, 7: number analyzed (Participants) | 8 | 7
  GSK2506102 (M5); 24 hours; n=8, 7 | NA (NA) — Mean and Standard Deviation were not calculable because concentration values were below detectable levels, but were imputed in the analysis. | NA (NA) — Mean and Standard Deviation were not calculable because concentration values were below detectable levels, but were imputed in the analysis.
  GSK2506104 (M3); 3 hours; n=8, 7: number analyzed (Participants) | 8 | 7
  GSK2506104 (M3); 3 hours; n=8, 7 | 0.2904 (0.02480) | 0.2938 (0.02618)
  GSK2506104 (M3); 12 hours; n=7, 7: number analyzed (Participants) | 7 | 7
  GSK2506104 (M3); 12 hours; n=7, 7 | 0.2970 (0.02959) | 0.2845 (0.02193)
  GSK2506104 (M3); 24 hours; n=6, 1: number analyzed (Participants) | 6 | 1
  GSK2506104 (M3); 24 hours; n=6, 1 | 0.3267 (0.03171) | 0.3016 (NA) — Data was not available as standard deviation could not be calculated for single participant.
  GSK2531398 (M6); 3 hours; n=8, 7: number analyzed (Participants) | 8 | 7
  GSK2531398 (M6); 3 hours; n=8, 7 | 0.2491 (0.02989) | 0.2444 (0.04833)
  GSK2531398 (M6); 12 hours; n=7, 7: number analyzed (Participants) | 7 | 7
  GSK2531398 (M6); 12 hours; n=7, 7 | 0.2500 (0.03259) | 0.2346 (0.02031)
  GSK2531398 (M6); 24 hours; n=8, 7: number analyzed (Participants) | 8 | 7
  GSK2531398 (M6); 24 hours; n=8, 7 | NA (NA) — Mean and Standard Deviation were not calculable because concentration values were below detectable levels, but were imputed in the analysis. | NA (NA) — Mean and Standard Deviation were not calculable because concentration values were below detectable levels, but were imputed in the analysis.
  GSK2531401 (M13); 3 hours; n=8, 7: number analyzed (Participants) | 8 | 7
  GSK2531401 (M13); 3 hours; n=8, 7 | 0.3595 (0.02324) | 0.3569 (0.03504)
  GSK2531401 (M13); 12 hours; n=7, 7: number analyzed (Participants) | 7 | 7
  GSK2531401 (M13); 12 hours; n=7, 7 | 0.3527 (0.03957) | 0.3386 (0.01580)
  GSK2531401 (M13); 24 hours; n=5, 1: number analyzed (Participants) | 5 | 1
  GSK2531401 (M13); 24 hours; n=5, 1 | 0.4154 (0.03151) | 0.3845 (NA) — Data was not available as standard deviation could not be calculated for single participant.

17. Secondary Outcome: Part 1: Maximum Observed Erythropoietin Concentration (Cmax, EPO) Following Administration of GSK1278863
Description: Venous blood samples were collected for measurement of plasma EPO at the indicated time points. Pharmacodynamic Population comprised of all participants in the Safety Population who had at least one pharmacodynamic assessment.
Time Frame: Pre-dose, 30 minutes, 1 hour, 1 hour 30 minutes, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 10 hours, 12 hours, 24 hours, 36 hours, and 48 hours post-dose
Population: Pharmacodynamic Population
Measure: Mean (Standard Deviation); unit: International units per liter
Arm/Group | Part 1: Moderate Hepatic Impairment Participants | Part 1: Healthy Participants
Number analyzed (Participants) | 8 | 8
International units per liter | 48.898 (36.8476) | 28.391 (13.1904)

18. Secondary Outcome: Part 2: Cmax, EPO Following Administration of GSK1278863
Description: Venous blood samples were collected for measurement of plasma EPO at the indicated time points following administration of GSK1278863.
Time Frame: as for outcome 17
Population: Pharmacodynamic Population
Measure: Mean (Standard Deviation); unit: International units per liter
Arm/Group | Part 2: Mild Hepatic Impairment Participants | Part 2: Healthy Participants
Number analyzed (Participants) | 12 | 9
International units per liter | 43.933 (20.2602) | 45.871 (35.1537)

19. Secondary Outcome: Part 1: Time of the Maximum Observed Erythropoietin Concentration (Tmax, EPO) Following Administration of GSK1278863
Description: as for outcome 18
Time Frame: as for outcome 17
Population: Pharmacodynamic Population
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 1: Moderate Hepatic Impairment Participants | Part 1: Healthy Participants
Number analyzed (Participants) | 8 | 8
Hours | 10.0 [8 to 12] | 10.0 [8 to 10]

20. Secondary Outcome: Part 2: Tmax, EPO Following Administration of GSK1278863
Description: as for outcome 18
Time Frame: as for outcome 17
Population: Pharmacodynamic Population
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 2: Mild Hepatic Impairment Participants | Part 2: Healthy Participants
Number analyzed (Participants) | 12 | 9
Hours | 10.0 [0 to 48] | 10.0 [6 to 12]

21. Secondary Outcome: Part 1: Erythropoietin Area Under the Concentration-time Curve From Time Zero (Pre-dose) to the Last Time of Quantifiable Concentration (AUC [0-t, EPO]) Following Administration of GSK1278863
Description: as for outcome 18
Time Frame: as for outcome 17
Population: Pharmacodynamic Population
Measure: Mean (Standard Deviation); unit: Hours* International units per liter
Arm/Group | Part 1: Moderate Hepatic Impairment Participants | Part 1: Healthy Participants
Number analyzed (Participants) | 8 | 8
Hours* International units per liter | 1262.3724 (1148.34702) | 697.7140 (393.05978)

22. Secondary Outcome: Part 2: AUC (0-t, EPO) Following Administration of GSK1278863
Description: as for outcome 18
Time Frame: as for outcome 17
Population: Pharmacodynamic Population
Measure: Mean (Standard Deviation); unit: Hours* International units per liter
Arm/Group | Part 2: Mild Hepatic Impairment Participants | Part 2: Healthy Participants
Number analyzed (Participants) | 12 | 9
Hours* International units per liter | 1258.6211 (683.32848) | 1061.7549 (647.67154)

23. Secondary Outcome: Part 1: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. A SAE is defined as any untoward medical occurrence that, at any dose that results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, is a congenital anomaly/birth defect or any other situation as per Medical or scientific judgment. Safety Population comprised of all participants who received at least one dose of study medication.
Time Frame: Up to 16 days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Moderate Hepatic Impairment Participants | Part 1: Healthy Participants
Number analyzed (Participants) | 8 | 8
Participants
  Any SAE | 0 | 0
  Any AE | 1 | 2

24. Secondary Outcome: Part 2: Number of Participants With AEs and SAEs
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. A SAE is defined as any untoward medical occurrence that, at any dose that results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, is a congenital anomaly/birth defect or any other situation as per Medical or scientific judgment.
Time Frame: Up to 16 days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Mild Hepatic Impairment Participants | Part 2: Healthy Participants
Number analyzed (Participants) | 12 | 9
Participants
  Any SAE | 0 | 0
  Any AE | 0 | 0

25. Secondary Outcome: Part 1: Number of Participants With Worst Case Hematology Results Relative to Potential Clinical Importance (PCI) Criteria Post-Baseline Relative to Baseline
Description: Blood samples were collected for analysis of hematocrit, hemoglobin, leukocytes, lymphocytes, neutrophils and platelets. PCI ranges were <0.075 or >0.54 proportion of red blood cells in blood for hematocrit, <25 or >180 grams per liter (g/L) for hemoglobin, <3 or >20 x10^9 cells per liter (cells/L) for leukocytes, <0.8 x10^9 cells/L for lymphocytes, <1.5 x10^9 cells/L for neutrophils, and <100 or >550 x10^9 cells/L for platelet. Participants were counted in worst case category that their value changes to (low, within range or no change or high), unless there is no change in their category. Participants whose laboratory value category was unchanged (example given [e.g.], High to High), or whose value became within range, were recorded in "To within Range or No Change" category. Participants were counted twice if the participant has values that changed 'To Low' and 'To High', so the percentages may not add to 100%. Baseline is defined as latest non-missing scheduled pre-dose assessment.
Time Frame: Baseline (Screening) and up to Day 16
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Moderate Hepatic Impairment Participants | Part 1: Healthy Participants
Number analyzed (Participants) | 8 | 8
Participants
  Hematocrit; To Low | 0 | 0
  Hematocrit; To within Range or No Change | 8 | 8
  Hematocrit; To High | 0 | 0
  Hemoglobin; To Low | 0 | 0
  Hemoglobin; To within Range or No Change | 8 | 8
  Hemoglobin; To High | 0 | 0
  Leukocytes; To Low | 1 | 0
  Leukocytes; To within Range or No Change | 7 | 8
  Leukocytes; To High | 0 | 0
  Lymphocytes; To Low | 0 | 0
  Lymphocytes; To within Range or No Change | 8 | 8
  Lymphocytes; To High | 0 | 0
  Neutrophils; To Low | 0 | 0
  Neutrophils; To within Range or No Change | 8 | 8
  Neutrophils; To High | 0 | 0
  Platelets; To Low | 0 | 0
  Platelets; To within Range or No Change | 8 | 8
  Platelets; To High | 0 | 0

26. Secondary Outcome: Part 2: Number of Participants With Worst Case Hematology Results Relative to PCI Criteria Post-Baseline Relative to Baseline
Description: Blood samples were collected for analysis of hematocrit, hemoglobin, leukocytes, lymphocytes, neutrophils and platelets. PCI ranges were <0.075 or >0.54 proportion of red blood cells in blood for hematocrit, <25 or >180 g/L for hemoglobin, <3 or >20 x10^9 cells/L for leukocytes, <0.8 x10^9 cells/L for lymphocytes, <1.5 x10^9 cells/L for neutrophils, and <100 or >550 x10^9 cells/L for platelet. Participants were counted in worst case category that their value changes to (low, within range or no change or high), unless there is no change in their category. Participants whose laboratory value category was unchanged (e.g., High to High), or whose value became within range, were recorded in "To within Range or No Change" category. Participants were counted twice if the participant has values that changed 'To Low' and 'To High', so the percentages may not add to 100%. Baseline is defined as latest non-missing scheduled pre-dose assessment.
Time Frame: Baseline (Screening) and up to Day 16
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Mild Hepatic Impairment Participants | Part 2: Healthy Participants
Number analyzed (Participants) | 12 | 9
Participants
  Hematocrit; To Low | 0 | 0
  Hematocrit; To within Range or No Change | 12 | 9
  Hematocrit; To High | 0 | 0
  Hemoglobin; To Low | 0 | 0
  Hemoglobin; To within Range or No Change | 12 | 9
  Hemoglobin; To High | 0 | 0
  Leukocytes; To Low | 0 | 0
  Leukocytes; To within Range or No Change | 12 | 9
  Leukocytes; To High | 0 | 0
  Lymphocytes; To Low | 1 | 0
  Lymphocytes; To within Range or No Change | 11 | 9
  Lymphocytes; To High | 0 | 0
  Neutrophils; To Low | 0 | 0
  Neutrophils; To within Range or No Change | 12 | 9
  Neutrophils; To High | 0 | 0
  Platelets; To Low | 0 | 0
  Platelets; To within Range or No Change | 12 | 9
  Platelets; To High | 0 | 0

27. Secondary Outcome: Part 1: Number of Participants With Worst Case Chemistry Results Relative to PCI Criteria Post-Baseline Relative to Baseline
Description: Blood samples were collected for analysis of following parameters. PCI ranges were <30g/L (albumin), <2 or >2.75 millimoles/L(mmol/L) (calcium), <3 or >9mmol/L(glucose), >=2 times Upper limit of Normal(ULN) units/L(U/L) (alanine aminotransferase [ALT]), >=2 times ULN U/L (alkaline phosphatase), >=2 times ULN U/L(aspartate aminotransferase [AST]), >=1.5 times ULN micromoles/L (µmol/L)(bilirubin), <3 or >5.5mmol/L(potassium), and <130 or >150mmol/L(sodium). Participants were counted in worst case category that their value changes to (low,within range or no change or high), unless there is no change in their category. Participants whose laboratory value category was unchanged (e.g., High to High), or whose value became within range, were recorded in To within Range or No Change category. Participants were counted twice if participant has values that changed To Low and To High, so the percentages may not add to 100%. Baseline is defined as latest non-missing scheduled pre-dose assessment.
Time Frame: Baseline (Screening) and up to Day 16
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Moderate Hepatic Impairment Participants | Part 1: Healthy Participants
Number analyzed (Participants) | 8 | 8
Participants
  ALT ; To Low | 0 | 0
  ALT;To within Range or No Change | 8 | 8
  ALT; To High | 0 | 0
  Albumin; To Low | 0 | 0
  Albumin; To within Range or No Change | 8 | 8
  Albumin; To High | 0 | 0
  Alkaline Phosphatase; To Low | 0 | 0
  Alkaline Phosphatase; To within Range or No Change | 8 | 8
  Alkaline Phosphatase; To High | 0 | 0
  AST; To Low | 0 | 0
  AST;To within Range or No Change | 8 | 8
  AST; To High | 0 | 0
  Bilirubin; To Low | 0 | 0
  Bilirubin; To within Range or No Change | 8 | 8
  Bilirubin; To High | 0 | 0
  Calcium; To Low | 0 | 0
  Calcium; To within Range or No Change | 8 | 8
  Calcium; To High | 0 | 0
  Glucose; To Low | 0 | 0
  Glucose; To within Range or No Change | 6 | 8
  Glucose; To High | 2 | 0
  Potassium; To Low | 0 | 0
  Potassium; To within Range or No Change | 8 | 8
  Potassium; To High | 0 | 0
  Sodium; To Low | 1 | 0
  Sodium; To within Range or No Change | 7 | 8
  Sodium; To High | 0 | 0

28. Secondary Outcome: Part 2: Number of Participants With Worst Case Chemistry Results Relative to PCI Criteria Post-Baseline Relative to Baseline
Description: Blood samples were collected for analysis of following parameters. PCI ranges were <30g/L (albumin), <2 or >2.75 mmol/L (calcium), <3 or >9mmol/L (glucose), >=2 times ULN U/L (ALT), >=2 times ULN U/L (alkaline phosphatase), >=2 times ULN U/L (AST), >=1.5 times ULN µmol/L (bilirubin), <3 or >5.5 mmol/L (potassium), and <130 or >150 mmol/L (sodium). Participants were counted in worst case category that their value changes to (low, within range or no change or high), unless there is no change in their category. Participants whose laboratory value category was unchanged (e.g., High to High), or whose value became within range, were recorded in To within Range or No Change category. Participants were counted twice if the participant has values that changed To Low and To High, so the percentages may not add to 100%. Baseline is defined as latest non-missing scheduled pre-dose assessment.
Time Frame: Baseline (Screening) and up to Day 16
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Mild Hepatic Impairment Participants | Part 2: Healthy Participants
Number analyzed (Participants) | 12 | 9
Participants
  ALT ; To Low | 0 | 0
  ALT;To within Range or No Change | 12 | 9
  ALT ; To High | 0 | 0
  Albumin; To Low | 0 | 0
  Albumin; To within Range or No Change | 12 | 9
  Albumin; To High | 0 | 0
  Alkaline Phosphatase; To Low | 0 | 0
  Alkaline Phosphatase; To within Range or No Change | 12 | 9
  Alkaline Phosphatase; To High | 0 | 0
  AST; To Low | 0 | 0
  AST;To within Range or No Change | 12 | 9
  AST; To High | 0 | 0
  Bilirubin; To Low | 0 | 0
  Bilirubin; To within Range or No Change | 12 | 9
  Bilirubin; To High | 0 | 0
  Calcium; To Low | 0 | 0
  Calcium; To within Range or No Change | 12 | 9
  Calcium; To High | 0 | 0
  Glucose; To Low | 0 | 0
  Glucose; To within Range or No Change | 10 | 9
  Glucose; To High | 2 | 0
  Potassium; To Low | 0 | 0
  Potassium; To within Range or No Change | 12 | 9
  Potassium; To High | 0 | 0
  Sodium; To Low | 0 | 0
  Sodium; To within Range or No Change | 12 | 9
  Sodium; To High | 0 | 0

29. Secondary Outcome: Part 1: Number of Participants With Abnormal Urinalysis Findings
Description: Urine samples were collected at indicated time points for the analysis of urine parameters including specific gravity and Potential of hydrogen (pH) of urine, presence of glucose, protein, blood, ketones, bilirubin, urobilinogen, nitrite, and leukocyte esterase in urine.
Time Frame: Up to Day 16
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Moderate Hepatic Impairment Participants | Part 1: Healthy Participants
Number analyzed (Participants) | 8 | 8
Participants | 0 | 0

30. Secondary Outcome: Part 2: Number of Participants With Abnormal Urinalysis Findings
Description: as for outcome 29
Time Frame: Up to Day 16
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Mild Hepatic Impairment Participants | Part 2: Healthy Participants
Number analyzed (Participants) | 12 | 9
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious adverse events (Non-SAEs) were collected from the start of the study treatment up to 16 days in each part of the study.
Description: SAEs and Non-SAEs were reported for Safety Population comprised of all participants who received at least one dose of study medication.
Arm/Group | Part 1: Moderate Hepatic Impairment Participants | Part 1: Healthy Participants | Part 2: Mild Hepatic Impairment Participants | Part 2: Healthy Participants
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/12 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/12 | 0/9
Other Adverse Events (participants affected / at risk) | 1/8 | 2/8 | 0/12 | 0/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Moderate Hepatic Impairment Participants (N=8) | Part 1: Healthy Participants (N=8) | Part 2: Mild Hepatic Impairment Participants (N=12) | Part 2: Healthy Participants (N=9)
Toothache (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-11-22): https://cdn.clinicaltrials.gov/large-docs/37/NCT03223337/SAP_000.pdf
  • Study Protocol (2017-05-23): https://cdn.clinicaltrials.gov/large-docs/37/NCT03223337/Prot_001.pdf